CLINICAL TRIAL: NCT04327960
Title: Risk Stratification in Pulmonary Embolism
Brief Title: Risk Assessment Strategies in Pulmonary Embolism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam louiz Azmy, Physician, Assiut University
Other Study IDs: Pulmonary embolism
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac troponin (cTn) — Cardiac troponin (cTn) will be measured with the Dimension RxL-HM analyzer .The one-step enzyme immunoassay is based on cTn specific monoclonal antibodies, performed on a separate module of the analyzer, assay-time is 17 minutes.

SUMMARY:
The aim of this study is to evaluate different scores of risk assessment in patients with pulmonary embolism. This study aim to compare the accuracy of these scores in predicting mortality during hospital admission.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a potentially life-threatening cardiovascular emergency with a high mortality rate.Approximately 1% of all hospitalized patients and 10% of all in-hospital mortalities are PE related. Adding to this, acute PE is linked to comparatively high (≥13%) short-term mortalities that occur either in hospital or within 30 days.

Some studies have demonstrated that PE may indicate increased 1-year mortality rates up to 25%,,. Therefore, PE is considered a potentially fatal disease, although patients who escape a PE-related death are still endangered by hematologic mishaps, especially recurrence of VTE and/or PE, or on the contrary, serious hemorrhage5.

Risk stratification of patients with acute PE is mandatory for determining the appropriate therapeutic management approach. Risk classification of PE can discriminate low-risk patients, who can be medicated as outpatients, from others at high risk, in whom a profit from intensive care unit admission or even in-hospital thrombolytic therapy is expected.

ELIGIBILITY:
Inclusion Criteria:

-

All patients will be subjected to the following:

1. Complete history taking and clinical examination.
2. Chest x-ray
3. ECG and echocardiography.
4. Arterial blood gases.
5. Multislice CT angiography of the chest.
6. Laboratory tests and biomarkers.

Exclusion Criteria:

* 1- Patients with unexpected or accidental diagnosis of PE (patients undergoing diagnostic tests for another suspected disease.

  2- Patients with acute left heart failure or acute respiratory failure responsible for symptoms.

  3- Patient with recurrent PE (only the first event was included in the analysis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study is a cross-sectional study. All patients consecutively admitted to Assuit University Hospital, diagnosid with PE will be included.
  At least 80 patients will be included in the present study. Sample size was calculated using Epi- Info version 7, based on a previous study conducted by Yousif and Hussein (2019), which demonstrated that the mortality rate from pulmonary embolism was 13.7%, with a confidence limit of 5% and a confidence level of 80%. To overcome the dropouts the sample may be extended to 100 patients.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary embolism-related death | Baseline
  Approximately 1% of all hospitalized patients and 10% of all in-hospital mortalities are PE related. Adding to this, acute PE is linked to comparatively high (≥13%) short-term mortalities that occur either in hospital or within 30 days

SECONDARY OUTCOMES:
hospital stay, need for ICU admission, need for mechanical ventilation or cardiopulmonary resuscitation or home dischage. | Baseline
  patients who escape a PE-related death are still endangered by hematologic mishaps, especially recurrence of VTE and/or PE, or on the contrary, serious hemorrhage

REFERENCES:
- [Background] Jimenez D, Lobo JL, Fernandez-Golfin C, Portillo AK, Nieto R, Lankeit M, Konstantinides S, Prandoni P, Muriel A, Yusen RD; PROTECT investigators. Effectiveness of prognosticating pulmonary embolism using the ESC algorithm and the Bova score. Thromb Haemost. 2016 Apr;115(4):827-34. doi: 10.1160/TH15-09-0761. Epub 2016 Jan 7. PMID 26738514
- [Background] Hobohm L, Hellenkamp K, Hasenfuss G, Munzel T, Konstantinides S, Lankeit M. Comparison of risk assessment strategies for not-high-risk pulmonary embolism. Eur Respir J. 2016 Apr;47(4):1170-8. doi: 10.1183/13993003.01605-2015. Epub 2016 Jan 7. PMID 26743479